CLINICAL TRIAL: NCT03258996
Title: Modified VISTA Technique Versus Coronally Advanced Flap in the Treatment of Class III Multiple Recessions: Randomized Clinical Trial
Brief Title: m-VISTA Technique vs. CAF in the Treatment of Class III Multiple Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aitziber Fernandez Jimenez (Other)
Responsible Party: Sponsor-Investigator, Aitziber Fernandez Jimenez, Principal Investigator, University of the Basque Country (UPV/EHU)
Organization: University of the Basque Country (UPV/EHU) (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017_01
Record Dates: First submitted 2017-08-18; First posted 2017-08-23 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Gingival Recessions
Keywords: Gingival recession; Class III gingival recession; Multiples gingival recessions; Periodontitis; Mucogingival surgery; Modified vestibular incision subperiosteal tunnel access; Coronally advanced flap; Connective tissue graft; Post-surgical pain
MeSH Terms: conditions — Gingival Recession; Periodontitis; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: We will perform the experimental or control technique according to the randomization sequence.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant: Initially, the subject will not know what technique has been received, the complete information regarding the surgical technique used, as the results obtained in his case, will be given in the last visit of the year.
  Observer: Another periodoncist (R.E.), outside the intervention, would be in charge of recording the clinical parameters.
  Analyst: The statistician (X.M.) does not know which treatment corresponds to each variable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified vestibular incision subperiosteal tunnel access (Experimental): Test group: Coverage of Class III multiples gingival recessions with the application of Modified vestibular incision subperiosteal tunnel access technique and a connective tissue graft from the palate.
  Interventions: Procedure: Modified vestibular incision subperiosteal tunnel access
- Coronally advanced flap (Active Comparator): Control group: Coverage of Class III multiples gingival recessions with the application of Coronally advanced flap and a connective tissue graft from the palate.
  Interventions: Procedure: Coronally advanced flap

INTERVENTIONS:
Procedure: Modified vestibular incision subperiosteal tunnel access — Single vertical mucosal incision, in the middel of the area to be treated, from which we began to lift a mucoperiosteal flap in a single plane.
  With a micro-scalpel intrasulcular incisions are made extending to the base of the papillas.
  Preparation of a tunnel in the same plane. Take a connective tissue graft on the same side of the palate. The connective graft is inserted through the vertical incision prepared with the aid of the suture.
  All is stabilized by means of suspensory sutures of coronal traction on each point of contact.
  Finally the vertical incision made is sutured.
  Other Names: m-VISTA
  Arms: Modified vestibular incision subperiosteal tunnel access
Procedure: Coronally advanced flap — Oblique submarginal incisions in both interdental areas of each recession, which continue with the intrasulcular incision, one tooth extending on each side of the teeth to be treated.
  A partial-total-partial thickness flap is elevated in the coronal-apical direction.
  A vestibular mucosal dissection is performed to eliminate muscle tension. The remnant tissue of the anatomical interdental papillas is desepithelized. Take a CTG on the same side of the palate. The connective tissue graft is stabilized with resorbable suture over the recessions with suspensory sutures on the teeth.
  Finally, suspensory sutures with non-resorbable sutures are also used to achieve an accurate adaptation of the vestibular flap over the exposed root and stabilize each surgical papilla over each desepithelized interdental area.
  Other Names: CAF
  Arms: Coronally advanced flap

SUMMARY:
The main objective is to assess whether the percentage of root coverage (%RC) achieved in the treatment of multiples class III recessions using the technique we have called modified vestibular incision subperiosteal tunnel access (m-VISTA), which is a lateral approach subperiosteal tunnel technique, combined with a connective tissue graft is greater than that achieved through the coronally advance flap (CAF) technique together with a connective tissue graft.

DETAILED DESCRIPTION:
The reason for designing this study is that treatment of Class III gingival recessions (Miller 1985) continues to be challenging today and, although different techniques have been proposed to attempt to improve root coverage results, there is little evidence on what would offer better results.

To achieve those objectives a randomized controlled clinical trial is designed. Using the percentage of root coverage as a primary response variable, it is estimated with the calculation of the sample size, we would need 11 patients for each treatment group (Domenech and Granero 2010). In addition, taking into account possible drop-outs, we would increase the number of patients by recruiting a total of 24 patients.

A same experienced, blind and calibrated (the intraclass correlation coefficient will be at least of 0.75) examiner (R.E.) will collect the following periodontal clinical parameters at the baseline, and at 6 and 12 months, in each tooth involved, using a periodontal probe: Gingival recession, number and location of recessions to be treated, number of treated recessions that have a complete root coverage, the width of the gingival recession and the keratinized gingiva, the distance from the contact point to the interdental papilla, depth of probing, bleeding index and plaque index. And will also collect the opinion of the participant regarding pain and the degree of satisfaction with the aesthetic result.

Students of the University of the Basque Country's (UPV/EHU) Own Degree in Periodontology and Osteointegration will perform the corresponding surgical technique (m-VISTA or CAF) depending on the randomization sequence obtained. A clinical monitor (A.M.G.) will keep the sequence hidden until the moment of the intervention.

Initially, the subject will not know which technique to receive, the complete information regarding the surgical technique used, as the results obtained in his case, will be given in the last visit of the year.

Finally, a blind statistic (X.M) will analyze the data using the SPSS software, having as unit of analysis the subject. Doing a descriptive statistics, checking if the groups are homogeneous in basal, inter-group, intra-group and change variables comparisons and logistical regression to assess the intensity and duration of post-surgical pain adjusted for possible confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the Master of Periodontology of the UPV / EHU.
* Age ≥ 18 years.
* Multiple recessions (more than two) Class III ≥ 2 mm deep, in which the interdental papilla does not extend beyond the cementoenamel line.
* Absence of active periodontal disease.
* Plaque index (O'Leary et al. 1972) and bleeding index (Ainamo and Bay 1975) ≤15%.
* Informed consent.

Exclusion Criteria:

* Smokers > 10 cigarettes / day.
* Subjects with systemic conditions that contraindicate surgery.
* Subjects that have taken analgesics and anti-inflammatory drugs in the last 72 hours.
* Subjects taking opioids, anticonvulsants and antidepressants except serotonin selective inhibitors.
* Women who are pregnant or nursing.
* Patients who do not wish to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of root coverage (%CR) | 12 months
  In each patient the mean of their gingival recessions at baseline (initial RECm) and at 12 months (RECm_12 months) will be calculated. A new variable called %CR [(RECm_initial - RECm_12 months) / (RECm_initial x 100) will be calculated.

SECONDARY OUTCOMES:
Percentage of recessions with complete root coverage (%CRC) | 12 months
  Each patient will record the number of recessions, which after treatment, show complete root coverage at 12 months (CRC_12 months). A new variable called % CRC_12 months [CRC_12meses / NRT x100] will be calculated.
Post-surgical pain perception | After surgery up to 14 days
  The subject will we instructed to collect their perception of post-surgical pain in the VAS based Journal of Pain (IDT). Specifically the subject will record: Its intensity (0-100mm), its duration (minutes or hours) and if any analgesic treatment has been necessary (No o Yes: Which?).
Gingival recession (REC) | Change from baseline at following surgery sixth and twelfth month respectively.
  Distance in mm from the amelocementaria line the gingival margin, measured at the vestibular midpoint. It will be registered in all the teeth present (except wisdom teeth) at the beginning, and, during the follow-up only in the recessions to be treated.
Post-surgical aesthetic result (VAS aesthetic) | 12 months
  The same examiner will evaluate the degree of satisfaction of the subject with the aesthetic result obtained after the intervention, through a Questionnaire based on the Visual Analogue Scale (VAS).
Pre-surgical pain perception | Baseline.
  In the VAS based Journal of Pain (IDT) the examiner will record if the subject has had regional head and neck pain in the last month and if there is any pain in the immediate preoperative, if it is affirmative the intensity will be noted.
Post-surgical complications | After surgery first seven days.
  The presence or not, as the description, of the post-surgical complications (PSC) that may appear will be collected.
Central Sensitization Inventory severity-level score of the subject | Baseline.
  Central Sensitization inventory (CSI) (Mayer et al. 2012) will be done, in which each subject will be asked on the frequency in which he perceives 25 symptoms and will be given a score of 0-4 finally establishing a clinical level in a range of 0-100 points (Subclinical: 0-29; Medium: 30-39; Moderate: 40-49 ; Severe: 50-59; Extreme: 60-100).
Number of recessions to be treated (NRT) Number of recessions to be treated (NRT) | Baseline.
  Number of Class III recessions to be treated will be recorded.
Localization of the recessions to treat (LRT) | Baseline.
  On the one hand, upper recessions will be considered the located in the maxillary and on the other hand, lower recessions those located in the mandible.
Gingival recession width (GRW) | Change from baseline at following surgery sixth and twelfth month respectively.
  Mesio-distal distance taken in the coronal area of the same, measured in millimeters. It will be recorded only in the recessions to be treated.
Keratinized gingiva width (KGW) | Change from baseline at following surgery sixth and twelfth month respectively.
  Distance in millimeters from the mucogingival junction to the gingival margin, measured at the vestibular midpoint. It will be recorded only in the recessions to be treated.
Distance from contact point to the interdental papilla (CP-IP) | Change from baseline at following surgery sixth and twelfth month respectively.
  Distance in millimeters from the mesial and distal contact point of the tooth with recession, to the most coronal part of the interdental papilla. It will be recorded only in the recessions to be treated.
Probing depth (PD) | Change from baseline at following surgery sixth and twelfth month respectively.
  Distance in millimeters from the gingival margin to the bottom of the periodontal pocket. It will be recorded at the beginning in all teeth present (except wisdow teeth) in 6 points per tooth (mesio-bucal, mid-bucal, disto-bucal, mesio-lingual, mid-lingual and disto-lingual) and, during follow-up, only in the recessions to be treated at the vestibular mid-point.
Patient bleeding index (BI) | Change from baseline at following surgery sixth and twelfth month respectively.
  After a periodontal probing of all teeth, the presence (yes or no) of bleeding is recorded dichotomously at 6 points per tooth (mesio-bucal, mid-bucal, disto-bucal, mesio-lingual, mid-lingual and disto-lingual) and the percentage of sites that bleed from the total of probed sites is calculated (Ainamo and Bay 1975).
Patient plaque index (PI) | Change from baseline at following surgery sixth and twelfth month respectively.
  A plaque developer is used and the presence (yes or no) of plaque is recorded dichotomously at 6 points per tooth (mesio-bucal, mid-bucal, disto-bucal, mesio-lingual, mid-lingual and disto-lingual) and the percentage of sites with plaque of the total probed sites is calculated (O'Leary et al 1972).

CONTACTS AND LOCATIONS:
Overall Officials: Luis Antonio Aguirre Zorzano, Dr., Study Director — University of the Basque Country (UPV/EHU); Aitziber Fernández Jiménez, Lcda., Principal Investigator — University of the Basque Country (UPV/EHU); Ruth Estefanía Fresco, Dr., Study Chair — University of the Basque Country (UPV/EHU); Xabier Marichalar Mendia, Dr., Study Chair — University of the Basque Country (UPV/EHU); Aroa Hereñu González, Lcda., Study Chair — University of the Basque Country (UPV/EHU); Jose Manuel Aguirre Urizar, Dr., Study Director — University of the Basque Country (UPV/EHU); Ana María García de la Fuente, Dr., Study Chair — University of the Basque Country (UPV/EHU)
Locations (1):
- Department fo Stomatology II, Faculty of Medicine and Nursery, University of the Basque Country, Leioa, Biscay, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data collected for the study will be identified by a code and only the researcher will be able to relate them. The personal data will be treated with absolute confidentiality in accordance with the Data Protection Law and will remain in the patient's clinical history. The coded data will be included in a UPV/EHU´s file with reference number 2080310015-INA0110, whose head is Ana María García de la Fuente, and will only be used for the purposes of this project.

REFERENCES:
- [Background] Agudio G, Nieri M, Rotundo R, Franceschi D, Cortellini P, Pini Prato GP. Periodontal conditions of sites treated with gingival-augmentation surgery compared to untreated contralateral homologous sites: a 10- to 27-year long-term study. J Periodontol. 2009 Sep;80(9):1399-405. doi: 10.1902/jop.2009.090122. PMID 19722789
- [Background] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834
- [Background] Armitage GC. Development of a classification system for periodontal diseases and conditions. Ann Periodontol. 1999 Dec;4(1):1-6. doi: 10.1902/annals.1999.4.1.1. PMID 10863370
- [Background] Aroca S, Keglevich T, Barbieri B, Gera I, Etienne D. Clinical evaluation of a modified coronally advanced flap alone or in combination with a platelet-rich fibrin membrane for the treatment of adjacent multiple gingival recessions: a 6-month study. J Periodontol. 2009 Feb;80(2):244-52. doi: 10.1902/jop.2009.080253. PMID 19186964
- [Background] Aroca S, Molnar B, Windisch P, Gera I, Salvi GE, Nikolidakis D, Sculean A. Treatment of multiple adjacent Miller class I and II gingival recessions with a Modified Coronally Advanced Tunnel (MCAT) technique and a collagen matrix or palatal connective tissue graft: a randomized, controlled clinical trial. J Clin Periodontol. 2013 Jul;40(7):713-20. doi: 10.1111/jcpe.12112. Epub 2013 Apr 30. PMID 23627374
- [Background] Butler BL. The subepithelial connective tissue graft with a vestibular releasing incision. J Periodontol. 2003 Jun;74(6):893-8. doi: 10.1902/jop.2003.74.6.893. PMID 12887003
- [Background] Carvalho PF, da Silva RC, Cury PR, Joly JC. Modified coronally advanced flap associated with a subepithelial connective tissue graft for the treatment of adjacent multiple gingival recessions. J Periodontol. 2006 Nov;77(11):1901-6. doi: 10.1902/jop.2006.050450. PMID 17076617
- [Background] Chatterjee A, Sharma E, Gundanavar G, Subbaiah SK. Treatment of multiple gingival recessions with vista technique: A case series. J Indian Soc Periodontol. 2015 Mar-Apr;19(2):232-5. doi: 10.4103/0972-124X.145836. PMID 26015680
- [Background] Daprile G, Gatto MR, Checchi L. The evolution of buccal gingival recessions in a student population: a 5-year follow-up. J Periodontol. 2007 Apr;78(4):611-4. doi: 10.1902/jop.2007.060277. PMID 17397306
- [Background] de Sanctis M, Zucchelli G. Coronally advanced flap: a modified surgical approach for isolated recession-type defects: three-year results. J Clin Periodontol. 2007 Mar;34(3):262-8. doi: 10.1111/j.1600-051X.2006.01039.x. PMID 17309597
- [Background] Del Corso M, Sammartino G, Dohan Ehrenfest DM. Re: "Clinical evaluation of a modified coronally advanced flap alone or in combination with a platelet-rich fibrin membrane for the treatment of adjacent multiple gingival recessions: a 6-month study". J Periodontol. 2009 Nov;80(11):1694-7; author reply 1697-9. doi: 10.1902/jop.2009.090253. PMID 19905939
- [Background] Kennedy JE, Bird WC, Palcanis KG, Dorfman HS. A longitudinal evaluation of varying widths of attached gingiva. J Clin Periodontol. 1985 Sep;12(8):667-75. doi: 10.1111/j.1600-051x.1985.tb00938.x. PMID 3902907
- [Background] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Background] Miller PD Jr. A classification of marginal tissue recession. Int J Periodontics Restorative Dent. 1985;5(2):8-13. No abstract available. PMID 3858267
- [Background] Molnar B, Aroca S, Keglevich T, Gera I, Windisch P, Stavropoulos A, Sculean A. Treatment of multiple adjacent Miller Class I and II gingival recessions with collagen matrix and the modified coronally advanced tunnel technique. Quintessence Int. 2013 Jan;44(1):17-24. doi: 10.3290/j.qi.a28739. PMID 23444157
- [Background] Muller HP, Eger T, Schorb A. Gingival dimensions after root coverage with free connective tissue grafts. J Clin Periodontol. 1998 May;25(5):424-30. doi: 10.1111/j.1600-051x.1998.tb02466.x. PMID 9650881
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- [Background] Pini-Prato GP, Cairo F, Nieri M, Franceschi D, Rotundo R, Cortellini P. Coronally advanced flap versus connective tissue graft in the treatment of multiple gingival recessions: a split-mouth study with a 5-year follow-up. J Clin Periodontol. 2010 Jul;37(7):644-50. doi: 10.1111/j.1600-051X.2010.01559.x. Epub 2010 May 11. PMID 20492074
- [Background] Santamaria MP, da Silva Feitosa D, Nociti FH Jr, Casati MZ, Sallum AW, Sallum EA. Cervical restoration and the amount of soft tissue coverage achieved by coronally advanced flap: a 2-year follow-up randomized-controlled clinical trial. J Clin Periodontol. 2009 May;36(5):434-41. doi: 10.1111/j.1600-051X.2009.01389.x. PMID 19419445
- [Background] Susin C, Haas AN, Oppermann RV, Haugejorden O, Albandar JM. Gingival recession: epidemiology and risk indicators in a representative urban Brazilian population. J Periodontol. 2004 Oct;75(10):1377-86. doi: 10.1902/jop.2004.75.10.1377. PMID 15562916
- [Background] Tatakis DN, Chambrone L, Allen EP, Langer B, McGuire MK, Richardson CR, Zabalegui I, Zadeh HH. Periodontal soft tissue root coverage procedures: a consensus report from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S52-5. doi: 10.1902/jop.2015.140376. Epub 2014 Oct 15. PMID 25315018
- [Background] Wennstrom JL. Mucogingival therapy. Ann Periodontol. 1996 Nov;1(1):671-701. doi: 10.1902/annals.1996.1.1.671. No abstract available. PMID 9118276
- [Result] Aroca S, Keglevich T, Nikolidakis D, Gera I, Nagy K, Azzi R, Etienne D. Treatment of class III multiple gingival recessions: a randomized-clinical trial. J Clin Periodontol. 2010 Jan;37(1):88-97. doi: 10.1111/j.1600-051X.2009.01492.x. Epub 2009 Nov 30. PMID 19968743
- [Result] Dandu SR, Murthy KR. Multiple Gingival Recession Defects Treated with Coronally Advanced Flap and Either the VISTA Technique Enhanced with GEM 21S or Periosteal Pedicle Graft: A 9-Month Clinical Study. Int J Periodontics Restorative Dent. 2016 Mar-Apr;36(2):231-7. doi: 10.11607/prd.2533. PMID 26901301
- [Result] Zadeh HH. Minimally invasive treatment of maxillary anterior gingival recession defects by vestibular incision subperiosteal tunnel access and platelet-derived growth factor BB. Int J Periodontics Restorative Dent. 2011 Nov-Dec;31(6):653-60. PMID 22140667
- [Result] Zucchelli G, De Sanctis M. Treatment of multiple recession-type defects in patients with esthetic demands. J Periodontol. 2000 Sep;71(9):1506-14. doi: 10.1902/jop.2000.71.9.1506. PMID 11022782
- [Derived] Fernandez-Jimenez A, Estefania-Fresco R, Garcia-De-La-Fuente AM, Marichalar-Mendia X, Aguirre-Urizar JM, Aguirre-Zorzano LA. Comparative study of the modified VISTA technique (m-VISTA) versus the coronally advanced flap (CAF) in the treatment of multiple Miller class III/RT2 recessions: a randomized clinical trial. Clin Oral Investig. 2023 Feb;27(2):505-517. doi: 10.1007/s00784-022-04746-w. Epub 2022 Oct 20. PMID 36264343
- [Derived] Fernandez-Jimenez A, Estefania-Fresco R, Garcia-De-La-Fuente AM, Marichalar-Mendia X, Aguirre-Zorzano LA. Description of the modified vestibular incision subperiosteal tunnel access (m-VISTA) technique in the treatment of multiple Miller class III gingival recessions: a case series. BMC Oral Health. 2021 Mar 20;21(1):142. doi: 10.1186/s12903-021-01511-5. PMID 33743644